CLINICAL TRIAL: NCT06922825
Title: Study Evaluating 68Ga-FAPI-46 Tumor Microenvironment Interaction in Solid Tumor Patients
Brief Title: Pilot Study Evaluating Tumor Microenvironment Interaction in Solid Tumor Patients
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No patients enrolled onto study. Administratively withdrawn.
Sponsor: Eben Rosenthal (Other)
Collaborators: Vanderbilt University Medical Center (Other); Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Sponsor-Investigator, Eben Rosenthal, Barry and Amy Baker Professor and Chair, Vanderbilt-Ingram Cancer Center
Organization: Vanderbilt-Ingram Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: VICCHN25009
Record Dates: First submitted 2025-04-03; First posted 2025-04-11 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor Cancer; Solid Tumor Malignancy; Cancer; Malignancy
Keywords: Immunotherapy; anti-body based therapy; abt; antibody based therapy; anti body based therapy; cancer; malignancy; solid tumor
MeSH Terms: conditions — Neoplasms | interventions — FAPI-46

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 68 Ga FAPI-46 (Experimental): Each participant who meets criteria will receive one dose of 68 Ga FAPI-46 via IV and then receive a whole body PET/CT Scan the same day of infusion. Participants will be asked to have a CT/MRI with contrast approximately one week after the study drug infusion and scan.
  Researchers will compare PET/CT images using 68Ga-FAPI-46 to compare uptake determined by MRI or CT with contrast as usual Standard of Care.
  Interventions: Drug: 68Ga-FAPI-46

INTERVENTIONS:
Drug: 68Ga-FAPI-46 — Participants will receive an IV injection of 68Ga-FAPI-46. Then, shortly after will undergo a PET/CT imaging using the 68Ga-FAPI-46. Additionally, MRI or contrast CT imaging will be conducted, either on the same day or within 14 days.

SUMMARY:
This pilot study aims to compare PET/CT imaging using 68Ga-FAPI-46 to imaging results from standard MRI or CT with contrast in patients with solid tumors undergoing biologic therapy. A total of 50 participants will receive an intravenous injection of 68Ga-FAPI-46 and undergo a PET/CT scan shortly after received the study drug. Imaging will occur before starting standard antibody-based therapy. Participants will then proceed with their treatment, and the study team will monitor them through chart reviews for up to 36 months to evaluate treatment response and any correlation with tumor uptake observed on PET/CT scans.

DETAILED DESCRIPTION:
This is a pilot study to compare PET/CT uptake of 68Ga-FAPI-46 to uptake parameters determined by Standard of Care MRI or CT with contrast. Patients with a solid tumor diagnosis who are scheduled to undergo biologic therapy will be included in the study. Following imaging, patients will begin standard of care antibody based therapy and standard of care follow-up.

This study is an open label, single institution, pilot study to determine if 68-Ga-FAPI-46 can predict tumor uptake in patients with solid tumor and if the 68-Ga-FAPI-46 uptake in the tumor positively correlates with response to antibody based therapies.

A total of 50 subjects will be enrolled in the study. Imaging will take place prior to initiation of treatment. Patients will then be administered an intravenous injection of 68-Ga-FAPI-46 after which subjects will undergo a PET/CT scan shortly after receiving the drug. Subjects will then undergo treatment as determined by their primary team. The study team will chart review subjects for 36 months ± 6 months with the possibility of extending this follow-up depending on immunotherapy treatment duration to extract treatment response information as documented by their primary treatment team.

Total duration of active participation per patient may last approximately 45 days.

The study will take around 84 ± 6 months from the time the study opens to accrual. The total duration per patient from time of enrollment to chart review is 36 ± 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19 years.
* Biopsy confirmed diagnosis of solid tumor malignancy scheduled to undergo antibody-based therapy
* Subjects diagnosed with any stage of disease who will undergo immunotherapy treatment.
* Have acceptable kidney function and clinical lab values.

Exclusion Criteria:

* Myocardial infarction (MI); cerebrovascular accident (CVA); uncontrolled congestive heart failure (CHF); significant liver disease; or unstable angina within 6 months prior to enrollment
* Females who are currently pregnant or breastfeeding
* Severe renal disease or anuria
* Inability to lie flat or remain still for the duration of the scan.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2027-01 (Estimated); Primary Completion 2032-04 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Determine the correlative relationship between 68Ga-FAPI-46 and tumor uptake. | Day 1 Scan to Day 15 Scan.
  PET/CT uptake of 68Ga-FAPI-46 will be compared to uptake parameters determined by MRI or CT with contrast.

SECONDARY OUTCOMES:
Assess the ability of 68Ga-FAPI-46 to predict response to ABT | Day 1 Scan to Day 30 follow up with physician
  PET/CT imaging with 68Ga-FAPI-46 agent administration (study drug) will be compared to predictive capability of conventional scoring systems (e.g., PD-L1 CPS) scoring from patient biopsy specimens (gold standard). Treatment response values will be determined by the patient's primary treatment team per standard of care assessment.
  The analysis is exploratory, intended to generate preliminary data for future studies. The proposed sample size is 50 subjects, with approximately two-thirds undergoing contrast-enhanced CT and one-third undergoing MRI. Based on simulations, the margin of error for a 95% confidence interval is expected to range from 0.13 to 0.26 for n = 37, depending on the true correlation (0.8 to 0.5), and from 0.21 to 0.37 for n = 13.

CONTACTS AND LOCATIONS:
Overall Officials: Eben Rosenthal, MD, Study Director — Vanderbilt University/Ingram Cancer Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot study, and the sample size is not designed to support confirmatory conclusions. The analysis is exploratory, intended to generate preliminary data for future studies.